CLINICAL TRIAL: NCT01028092
Title: mTor-inhibitor (EVERolimus) Based Immunosuppressive Strategies for CNI Minimisation in OLD for Old Renal Transplantation
Acronym: EVEROLD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Novartis (Industry); Roche Pharma AG (Industry); Genzyme, a Sanofi Company (Industry); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVEROLD; RB 09.074
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Renal Transplant
MeSH Terms: interventions — Cyclosporine; thymoglobulin; Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (Active Comparator): anti R-IL2 induction + Mycophenolate Mofetil + cyclosporine A + corticosteroids
  Interventions: Drug: Anti R-IL2 + Cyclosporine
- CNI-free (Experimental): Thymoglobulin + Mycophenolate Mofetil + everolimus + corticosteroids
  Interventions: Drug: Thymoglobulin + Everolimus
- Switch (Experimental): anti R-IL2 + Mycophenolate Mofetil + (Cyclosporine then Everolimus) + corticosteroids
  Interventions: Drug: Anti R-IL2 + Cyclosporine then Everolimus

INTERVENTIONS:
Drug: Anti R-IL2 + Cyclosporine — * anti R-IL2 induction (Simulect ®, 20 mg D0 and D4)
  * Mycophenolate Mofetil (Cellcept ®) 3 grams per day beginning at D0
  * cyclosporine A (Neoral ®) started from 6 to 8 mg/kg adjusted to C2
  * corticosteroids 250 mg IV before and after surgery, then 1 mg/kg one week and 20mg/j the week after, then tapered until 10 mg/j at M1, 5 mg at M3 and stop between M4 and M6
  Arms: Control
Drug: Thymoglobulin + Everolimus — * Thymoglobulin ® induction started at 1.5mg/kg/j then adjusted to CD2 or total lymphocytes count, for 5 days
  * Mycophenolate Mofetil (Cellcept ®) 3 grams per day beginning at D0
  * everolimus (Certican ®): 4 to 6 mg/day started at D5, adjusted to achieve a residual level between 6 et 10 ng/ml
  * corticosteroids 250 mg IV before and after surgery, then 1 mg/kg one week and 20mg/j the week after, then tapered until 10 mg/j at M1, 5 mg at M3 and stop between M4 and M6
  Arms: CNI-free
Drug: Anti R-IL2 + Cyclosporine then Everolimus — * anti R-IL2 induction (Simulect ®, 20 mg D0 and D4)
  * Mycophenolate Mofetil (Cellcept ®) 3 g/d beginning at D0
  * cyclosporine A (Neoral ®) beginning at 6 to 8 mg/kg adjusted to C2, then switch to everolimus (Certican ®) between at W6, started at 3 mg/d, then adjusted to achieve a residual level between 6 et 10 ng/ml
  * corticosteroids 250 mg IV before and after surgery, then 1 mg/kg one week and 20mg/j the week after, then tapered until 10 mg/j at M1, 5 mg at M3 and stop between M4 and M6
  Arms: Switch

SUMMARY:
This study is designed to evaluate efficacity and safety of everolimus or (cyclosporine then everolimus) vs. cyclosporine as immunosuppressive treatment in renal transplantation for elderly (>60 years old) recipients receiving graft from elderly donor(>60 years old).

ELIGIBILITY:
Inclusion Criteria:

* Patient who has given written informed consent to participate in the study
* First or second single transplantation of a recipient (male or female) older than 60 years old
* Donor older than 60 years old
* PRA < 30%

Exclusion Criteria:

* Living donor
* Third transplantation
* PRA > 30%

Other protocol-defined inclusion/exclusion criteria may apply.

* Recipient of multi-organ transplant
* Active major infections (HBV, HCV, HIV)
* Loss of a first graft for immunologic issues
* Anemia (<9g/l) or leucopenia (<2500/mm3)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 327 (Actual)
Dates: Start 2009-03; Primary Completion 2014-03 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
calculated renal function with MDRD equation | 12 months

SECONDARY OUTCOMES:
Acute rejection rate | 12 months
Patient and graft survival rate | 12 months
Adverse events | 12 months
GFR calculated with Cockcroft Gault formula | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE MEUR, MD/PhD, Principal Investigator — CHU de Brest
Locations (18):
- France (18):
  - CHU Amiens, Amiens
  - CHU Pellegrin - Bordeaux, Bordeaux
  - CHRU de BREST, Brest
  - CHU Cote de Nacre, Caen
  - CHU Clermont Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Montpellier, Montpellier
  - CHU Nice, Nice
  - AP-HP Hopital Necker, Paris
  - CHU Poitiers, Poitiers
  - CHU Reims, Reims
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - Hopitaux Universitaires de Strasbourg, Strasbourg
  - CHU Rangueil - Toulouse, Toulouse
  - CHU Tours, Tours